CLINICAL TRIAL: NCT04370821
Title: COVID-19 CHAMPS Study of Healthcare, First Responder and Service Workers
Acronym: CHAMPS
Status: Active, not recruiting | Type: Observational
Sponsor: Villanova University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB FY2020-215
Record Dates: First submitted 2020-04-27; First posted 2020-05-01 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Occupational Exposure to SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The COVID-19 CHAMPS Study will obtain data on the physical and mental health and well-being of workers potentially exposed to the SARS-CoV-2 virus in the course of their duties. Included are a broad range of occupations including those working in the community (police officers, firefighters, emergency personnel, screening staff) as well as in permanent or temporary sites that care for patients (service staff, nurses, physicians and other health professionals). CHAMPS will obtain data on various exposure factors and health and create a registry of participants for extended follow up and sub-studies.

DETAILED DESCRIPTION:
The objective of the US COVID-19 CHAMPS Study is to assess the short- and long-term physical, social and behavioral health of all who were involved in supporting or delivering care for COVID-19 patients. Included are first responders, maintenance and support staff as well as healthcare professionals of all specialties and services. Initially the study will obtain data on the working environment and emotional and physical health. Additional data will be obtained on self-management, response strategies, effects on family, social and personal life and careers. This well-characterized cohort of workers will enable characterization of the health and social effects of their service, and prospective research on their future physical and mental health. It will also serve as a registry for future, hypothesis-driven sub-studies of behavioral and biological coping mechanisms and allostatic load, as well as randomized clinical trials. Participants will be recruited throughout the United States and its territories (Puerto Rico, Guam, the US Virgin Islands) with outcomes followed longitudinally for twenty years.

Initial analysis will be descriptive and include computation of frequency distributions, adjusted odds ratios and 95% confidence intervals. Multiple logistic regression methods will be used to assess association of health symptoms or conditions with estimates of exposure to COVID-19. Psychological distress will be estimated from self-reported responses to validated psychological instruments and survey items created to capture the unique aspects of exposure to COVID-19 in workplace settings. Odds rations will be adjusted for sex, age, race/ethnicity and job classification. The logistic regression model(s) will include self-reported baseline health status and other variables. Preliminary explorations of variable associations will be performed to aid with the development of sub-studies from the registry.

No direct health benefits are anticipated for participating in the study, but participants may learn about their health. Participation in the study provides the participants the opportunity to express the impact of responding to the COVID-19 pandemic on their health, which may be a source of relief. Participants may feel satisfaction about sharing information about their experiences that may help healthcare systems to plan for future health-related emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Working in a facility that screens, diagnoses, or treats COVID-19 patients or in the community as a first responder.
* Able to read and speak English

Exclusion Criteria:

* Anyone not meeting Inclusion Criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any adult exposed to increased risk of infection by SARS-CoV-2 as a result of work in the community or in settings where COVID-19 patients are screened, diagnosed or receive care. Included are first responders (e.g., police officers, firefighters, emergency medical technicians, paramedics) service employees (office staff, maintenance, housekeeping, food service), and healthcare professionals (e.g., physicians, nurses, phlebotomists, respiratory therapists, pharmacists).
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Estimated)
Dates: Start 2020-05-09 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Sample Size of enrolled CHAMPS Study participants by demographic characteristics during the first two years of the study | Two years
Exposure to SARS-CoV-2 based on models computed from participant baseline data and community variables, if available. | Two years
Infectious disease and chronic disease incidence rates by demographic characteristics | Four years
Completeness of data by demographic characteristics. | Two years

SECONDARY OUTCOMES:
Participation rates in ancillary and sub-studies within the CHAMPS registry. | four years
Number of participants enrolled in randomized trials based on the CHAMPS registry | four years

CONTACTS AND LOCATIONS:
Overall Officials: Heather Brom, PhD, Principal Investigator — Villanova University; Donna Havens, PhD,RN,FAAN, Principal Investigator — Villanova University
Locations (1):
- Villanova University, Villanova, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaufmann PG, Havens DS, Mensinger JL, Bradley PK, Brom HM, Copel LC, Costello A, D'Annunzio C, Dean Durning J, Maldonado L, Barrow McKenzie A, Smeltzer SC, Yost J; CHAMPS Study Investigators. The COVID-19 Study of Healthcare and Support Personnel (CHAMPS): Protocol for a Longitudinal Observational Study. JMIR Res Protoc. 2021 Oct 7;10(10):e30757. doi: 10.2196/30757. PMID 34582354